CLINICAL TRIAL: NCT00051688
Title: Tezacitabine and Oxaliplatin for the Treatment of Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Chiron Corporation (Industry)
Purpose: Treatment
Other Study IDs: TEZ101
Record Dates: First submitted 2003-01-15; First posted 2003-01-16 (Estimated); Last update posted 2006-07-11 (Estimated); Status verified 2006-07

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tezacitabine; Oxaliplatin

INTERVENTIONS:
Drug: tezacitabine
Drug: oxaliplatin

SUMMARY:
The primary purpose of this study is to determine the best dose of tezacitabine when combined with oxaliplatin in patients with metastatic colorectal cancer. This study will also evaluate tumor response to the combination of anti-cancer drugs.

ELIGIBILITY:
* Patients with metastatic colorectal adenocarcinoma who have failed one prior course of chemotherapy.
* Patients must have at least one measurable tumor.
* Patients may not have received prior treatment with oxaliplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - ACRC/Arizona Clinical Research Center, Tucson, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Cancer Institute Medical Group, Santa Monica, California
  - Georgetown University Medical Center, Lombardi Cancer Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Kansas City Oncology and Hematology Group, Kansas City, Missouri